CLINICAL TRIAL: NCT00840164
Title: Pathology of Skin, Nerve and Vasculature in the Amputated Limb of Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200812048R
Record Dates: First submitted 2009-02-08; First posted 2009-02-10 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-08

CONDITIONS: Wound; Diabetes; Amputation
Keywords: small-fiber sensory neuropathy; nerve pathology; vasculature pathology; amputation; diabetic foot wound; sensory neuropathy; below knee amputation
MeSH Terms: conditions — Wounds and Injuries; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — After amputation, sural nerve, posterior tibial nerve, and the accompanying vasculature will be harvested from the amputated leg. 3mm-puch skin will be taken from the amputated leg, 10 cm above the lateral malleolus.
Oversight: Data Monitoring Committee: No

SUMMARY:
1. To explore the pathology of nerve, vascular, and skin in the amputated leg
2. To diagnose small-fiber sensory neuropathy of the contralateral leg by investigating the skin intervention
3. To search for (1) mechanisms of amputation and (2) prevention measures for further amputation in the currently healthy-looking limb

DETAILED DESCRIPTION:
Diabetic foot occurs in 15% of diabetic population (3) and 15% of the diabetic foot patients end up with lower limb amputation. Peripheral neuropathy (sensory, motor and autonomic), peripheral vascular disease, trauma, infection and poor wound healing all contribute to diabetic foot problem.

Peripheral neuropathy could be evaluated in a variety of ways, including vibratory thresholds, thermal thresholds, pressure perception thresholds, muscle strength. All these predict foot ulceration to some degree(1). Motor nerve conduction velocity is an independent predictor for the development of new foot ulcer in diabetic population.

For more detailed structural study of neuropathy in diabetic patient, we could use skin biopsy method. Skin biopsy with PGP9.5 immunohistochemistry has been demonstrated by ultrastructural studies to label the terminal portions of both small myelinated and unmyelinated nerve in the epidermis . Intra-epidermal nerve fiber (IENF) density is reduced in patient with impaired glucose tolerance and clinically overt diabetes . Previous IENF density study was performed in diabetic patients with sensory symptom but no foot ulcer. Now we tried to evaluate IENF density in severe diabetic foot patient who received below knee amputation. Skin biopsy willl be performed at amputated leg. The skin biopsy area will be located at lateral side of distal leg, 10 cm above the lateral malleolus as previous protocol of our group . Underlying sural nerve and posterior tibial nerve will be also harvested for further ultra-structural study. The result will be compared to the control group which were recruited from a previously described cohort matched by gender and age.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic foot wound patient who underwent below-knee amputation

Exclusion Criteria:

* Diabetic foot wound patient who couldn't receive below-knee amputation due to severe heart disease, high anesthetic risk.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetic foot wound patient who underwent below-knee amputation due to poor wound healing and severe infection condition. The patient population often receives leg revasculariztion surgery but poor response for wound healing.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hsien Hsieh, Principal Investigator — Plasty surgery department, National Taiwan University Hospital
Locations (1):
- Plasty surgery department, National Taiwan University Hospital, Taipei, Taiwan